CLINICAL TRIAL: NCT06748716
Title: Effect of Blue Light Blocking on Reducing Manic Symptoms in Bipolar Disorder: a Randomized Placebo-controlled Trial BLUME (Blue Light Filtering in Manic Episodes)
Brief Title: Effect of Blue Light Blocking on Reducing Manic Symptoms in Bipolar Disorder
Acronym: BLUME
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rayan NASSERDINE (Other)
Responsible Party: Sponsor-Investigator, Rayan NASSERDINE, Associated investigator, Medical Doctor, Clinical chef in HUG, Department of psychiatry, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRD 17-2024-II
Record Dates: First submitted 2024-12-06; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Bipolar; Manic; Bipolar Disorder (BD); Dark Therapy; Actigraphy; Mania; RCT; Virtual Darkness
MeSH Terms: conditions — Mania; Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clear glasses (Placebo Comparator)
  Interventions: Device: Clear glasses
- Orange glasses (Experimental): Intervention group
  Interventions: Device: Blue-blocking glasses

INTERVENTIONS:
Device: Blue-blocking glasses — The investigators hypothesize that blue-blocking glasses (intervention) is more effective than placebo.
  Arms: Orange glasses
Device: Clear glasses — Clear-lensed glasses are placebo
  Arms: Clear glasses

SUMMARY:
This study will be a randomized controlled trial (RCT) measuring the efficacy of wearing blue-blocking glasses (orange glasses) on manic symptoms in a population of patients suffering from Bipolar Disorder (BD), hospitalized for a manic episode on 10 days compared to non-filtering glasses (clear glasses, placebo) in addition to pharmacological treatment as usual.

The primary objective of this study is to evaluate the efficacity of orange glasses on improving manic symptoms in adult patients presenting BD in comparison with placebo. The primary outcome will be the change of total score of the Young Mania Rating Scale (YMRS) from baseline to day 10. Secondary objectives will be change in sleep quality, in motor activity (patterns of activity and rest), impact on psychotics symptoms, kinetics of the decrease of the manic symptoms from inclusion to the study and impact on maximal administered antipsychotic medication dosage ; they will be explored.

The investigators hypothesize that orange glasses is more effective than placebo in improving manic symptoms as an adjuvant treatment.

This project will take place in Alizé unit which is a newly conceived specialized ward dedicated to treating BD, at the HUG. The methodology has been developed in collaboration with the center of clinical research (CRC). The study will be conducted in accordance with established ethical and data management/protection practices.

DETAILED DESCRIPTION:
The design of the study is a monocentric, single-blinded, two-arm parallel-group randomized placebo-controlled trial in a newly developed specialized mood disorder ward at the Geneva University Hospitals. The methodological aspects of this trial are elaborated in consultation with the Centre of Clinical Research (CRC) of our Hospital. The adjunctive treatment consists in wearing BBG for a few hours between 7pm and bedtime for ten days. Orange glasses (intervention) are from Melamedic®, type UV530 (Medical Device Class I - 93/42 EEC made in Denmark).

The adjunctive treatment will be compared to a placebo (clear-lensed glasses), both groups will also receive an active treatment as usual (the standard of care for treating manic episode following Swiss and international guidelines). No treatments are prohibited. All pharmacological treatments will be recorded. Due to the particularity of the device, the clinicians and the patient cannot be blind to the treatment condition (orange glasses vs clear glasses) which is an acknowledged limitation. The participants were masked to group assignment by receiving identical limited information about the purpose of the study : testing the effectiveness of different types of glasses in reducing manic symptoms by blocking different wavelengths of light. Patients will be randomized after eligibility has been established and written consent has been sought. If the patient capacity to consent is impaired, legal representative will be informed and capacity to consent will be re-assessed before each visit to obtain a written consent (delayed consent). Signs showing that the participant is unwilling to participate in the study will result in the participant exclusion (explicit refusal). The expected total duration of participation is 10 days. Data will be analyzed in an intention-to-treat design.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized with manic symptoms in HUG
* Diagnostic of Bipolar Disorder according to the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) criteria
* aged 18-70 years

Exclusion Criteria:

* previous knowledge of blue-blocking glasses
* not consenting to participate
* severe eye disease or traumatic injury affecting both eyes.
* withdrawal symptoms from any drug or alcohol at the time of admission (the start of the intervention will be delayed until withdrawal symptoms have ceased)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Manics symptoms | from baseline to day 10
  The primary endpoint will be the change of total score of the Young Mania Rating Scale (YMRS) from baseline to day 10. The YMRS is a checklist of 11 items that are ranked on a scale of 0-4 or 0-8, the latter anchoring given to the four items which can be rated even with patients with poor cooperation. The score range therefore is between 0 and 60. This scale is classically used to assess the effectiveness of the treatment on manic symptoms. This is a clinical interview scale to assess the severity of manic states primarily used for research and it is designed to measure the severity of manic states, it can help guide clinicians on treatment planning and progress.
  The investigators define a score of at least 20 points on the YMRS (> 20) to identify a manic state and the lower the score, the more the patient is in a state of euthymia (scale <2).

SECONDARY OUTCOMES:
Sleep quality | from baseline to day 10
  The investigators aim to assess the sleep quality for each participant by the Pittsburgh Sleep Quality Index (PSQI) and hypothesize that the patients receiving the intervention will have a better sleep quality.
  The scale assesses a broad range of sleep domains and consists of 19 self-rated questions that measure seven components of sleep that are scored from 0 to 3: sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleep medication and daytime dysfunction. The global score is the combination of the seven sub-scores and ranges therefore from 0 to 21, with higher scores for worse sleep quality; the cut-off point to define "poor sleepers" is >5.
Psychotics symptoms | from baseline to day 10
  The investigators aim to assess the presence or absence of psychotics symptoms by the Positive and Negative Syndrome Scale (PANSS).
  The scale has mostly been used to inventory, grade and follow the symptoms in schizophrenia. It quantifies positive symptoms, which refer to an excess or distortion of normal functions (e.g., hallucinations and delusions), and negative symptoms, which represent a diminution or loss of normal functions. The PANSS is composed of 3 subscales: Positive Scale, Negative Scale, and General Psychopathology Scale. Each subscale is rated with 1 to 7 points ranging from absent to extreme. The range for the Positive and Negative Scales is 7-49, and the range for the General Psychopathology Scale is 16-112
Kinectics of the decrease of manics symptoms | from baseline to day 10
  The investigators aim to assess the kinetics of the decrease of manics symptoms for each participtant and hypothesize that participants receiving the intervention will have a faster decrease in the Young Mania Rating Scale (YMRS).
Impact on maximal administred antipsychotic medication dosage | from baseline to day 10
  The investigators aim to record the dosage of antipsychotic treatment for each patient and hypothesize that participants receiving the intervention will have lower dosage.
Measure of the motor activity | from baseline to day 10
  The investigators aim to assess the intensity of the motor activity for each participant by actigraphy which is a noninvasive technique that measures physical activity levels of a subject by means of a wristwatch-like motion-sensing device that can be worn for prolonged periods of time. By use of a wrist-worn actigraph, motor activity will be continuously recorded for all groups.
  They will be compared to data from a healthy control group.

OTHER OUTCOMES:
Depressive symptoms | from baseline to day 10
  The investigators aim to assess the incidence and severity of depressive symptoms (in manic episode) or aggravation of depressive symptoms (in manic episode with mixed features) by the Montgomery-Asberg Depression Rating Scale (MADRS). The rating should be based on a clinical interview moving from broadly phrased questions about symptoms to more detailed ones which allow a precise rating of severity. Each item has a severity scale from 0 to 6, with higher scores reflecting more severe symptoms. Ratings can be added to form an overall score (from 0 to 60). This is our cut-offs : scores of 0-6 indicate an absence of symptoms; 7-19 represent mild depression; 20-34 moderate; 35-60 indicate severe depression.
Side effects | from baseline to day 10
  All adverse effects will be rigorously monitored during the whole study for each participant.
  Number of participants with treatment-related adverse events will be recorded if present.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopitaux Universitaires de Genève, Geneva, Suisse, Switzerland

IPD SHARING:
Plan to Share IPD: No